CLINICAL TRIAL: NCT05203770
Title: Adaptations of the Brain in Chronic Pain With Opioid Exposure I
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Principal Investigator, Northwestern University
Other Study IDs: STU00207384
Record Dates: First submitted 2021-11-16; First posted 2022-01-24 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Chronic Back Pain; Opioid Use
Keywords: Opioids; Opioid Misuse Disorder; Brain Adaptations; biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CBP+mOUD: Chronic Back pain participants taking opioids and classified in the opioid misuse disorder group
- CBP+O: Chronic Back pain participants taking opioids and without opioid misuse disorder group
- CBP-O: Chronic Back pain participants not taking opioids
- Healthy Controls: Healthy control without pain or taking opioids.

SUMMARY:
This study investigates brain reorganization and behavioral responses in chronic pain with opioid exposure in Chronic Back Pain (CBP).

DETAILED DESCRIPTION:
Chronic back pain (CBP) is the most prevalent chronic pain condition in the US. Opiates are commonly prescribed to treat CBP; as such, these patients are a primary contributor to the current opioid epidemic. This study will assess the impact of opioid use on brain anatomy and function in those subjects taking opioids without opioid misuse disorder, as well as those subjects with opioid misuse disorder, relative to those with CBP and are not taking opioids and healthy controls. This is an observational study, that seeks to establish risk factors and brain biomarkers for opioid misuse disorder and relate brain adaptations to exposure to both opioids and chronic pain. This study also seeks to determine the impact of opioid use on cognitive, emotional, and motor abilities.

ELIGIBILITY:
Inclusion Criteria:

* History of low back pain for a minimum of 6 months daily (prior to screening), meeting the Quebec Task Force Classification System symptom categories I-III;
* Male or female, age equal or greater than 18 years, with no racial/ethnic restrictions;
* Must have a Visual Analog Scale (VAS) pain score ≥ 40 mm (of 100 mm maximum) at the baseline scanning visit (for which 0mm = no pain, and 100 mm = worst pain imaginable);
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires;
* Must be in generally stable health;
* Must sign an informed consent document after a complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits and potential risks, and are willing to participate;
* Must have, on average ≥ 4/10 units of pain intensity over the course of a 1-2 week period prior to the brain scanning visit;
* Must be willing to complete daily smartphone/computer app ratings;
* Must be on regular opioid or NSAID therapy for at least 3 months prior to randomization (for opioid and non-opioid treatment groups, respectively), which will be up to the clinical investigator's decision.

Exclusion Criteria:

* Low back pain associated with any systemic signs or symptoms, e.g., fever, chills;
* Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures,
* fibromyalgia, history of tumor in the back;
* Other comorbid chronic pain or neurological conditions;
* Involvement in litigation regarding their back pain or having a disability claim or receiving workman's compensation or seeking either as a result of back pain;
* Diagnosis of current major depression or psychiatric disorder requiring treatment, or such a diagnosis in the previous 6 months;
* Beck Depression Inventory II score of >28;
* Use of therapeutic doses of antidepressant medications at unstable doses (i.e., tricyclic depressants,
* SSRIs, SNRIs; low doses used for sleep may be allowed);
* Significant other medical disease such as diabetes, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy;
* Uncontrolled hypertension;
* Renal insufficiency;
* Current use of recreational drugs or history of alcohol or drug abuse;
* Any change in medication for back pain in the last 30 days;
* High dose opioid prophylaxis, as defined as > 50mg morphine equivalent/day;
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Evidence of poor treatment compliance, in the judgment of the investigator;
* Intra-axial implants (e.g. spinal cord stimulators or pumps);
* All exclusion criteria for MR safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia;
* Pregnancy, or inability to use an effective form of contraception in women of child-bearing age;
* Diabetes (type 1 or type 2);
* Lactose intolerance;
* Allergic reaction to naproxen or any NSAID;
* Any untoward reaction to l-dopa or carbidopa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must be 18 years or older. Male and Female No racial/ethnic restrictions General health status: generally good health
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine effects of opioid exposure on human brain anatomy and function in CBP using resting-state functional magnetic resonance (fMRI). | 1-2 years
  We will test the impact of opioid use on brain anatomy and function. For this, all participants will undergo a resting-state functional magnetic resonance (fMRI) exam. Measures of brain anatomy and brain connectivity will be acquired and compared between the observational groups (CBP+O and CBP+mOUD, relative to CBP-O and healthy control). We seek to establish risk factors and brain biomarkers for OUD and relate brain adaptations to exposure to both opioids and chronic pain.
To determine cognition, emotion, and motor abilities with opioid exposure in CBP, and to identify associated human brain maladptions. | 1-2 years
  We will test the impact of opioid use on abilities in CBP+O and CBP+mOUD, relative to CBP-O and healthy controls. For this participants will respond to questionnaires related to their thoughts and feelings.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Shirley Ryan Ability Lab, Chicago, Illinois